CLINICAL TRIAL: NCT07344519
Title: Open-Label, Dose Escalation Early Phase 1 Study of ER2001 Intravenous Injection Repetitive Treatment in Adults With Early Manifest Huntington's Disease.
Brief Title: The Safety and Tolerability Study With ER2001 Intravenous Injection Repetitive Treatment in Adults With Early Manifest Huntington's Disease.
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: ExoRNA Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ER2001-002
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-01

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Intervention Model Description: As designed, the single group will be divided into 3 cohorts. The planned increasing doses are 0.08, 0.16, and 0.32 mg/kg, respectively in subsequent. If the safety is confirmed and decision made to proceed to the next higher dose, the next cohort of 3 participants will receive a higher dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ER2001 Injection (Experimental): The minimum initial dose is 0.08mg/kg, then escalate to 0.16mg/kg, and 0.32mg/kg. The planned duration of the treatment is 6 weeks, and ER2001 will be administrated intravenously at the first day of weeks 1, 2, 3, 4, 5, and 6.
  Interventions: Drug: ER2001 injection

INTERVENTIONS:
Drug: ER2001 injection — The minimum initial dose is 0.08mg/kg, then escalate to 0.16mg/kg, and 0.32mg/kg. The planned duration of the treatment is 6 weeks, and ER2001 will be administrated intravenously at the first day of weeks 1, 2, 3, 4, 5, and 6.

SUMMARY:
This is an open label, dose escalation clinic trial to evaluate safety, tolerability and pharmacokinetics with ER2001 Intravenous Injection repetitive treatment in Huntington's Disease patients who Completed Study ER2001-001（NCT06024265）. Furthermore, pharmacodynamics in particular target engagement, and clinical signs of efficacy will be assessed. This study will evaluate increasing doses of ER2001 in sequential cohorts. ER2001 was escalated over 3 dose levels . The planned duration of this additional treatment is 6 weeks for one course.

DETAILED DESCRIPTION:
The study include a screening period (4 week prior to the first administration), a treatment period (for 6 consecutive weeks, once a week [QW] for 6 weeks), and a safety follow-up period (12 weeks). Participants will receive 6 injections at the same dose level used in the NCT06024265 study, once a week over a period of 6 consecutive weeks. Planned doses for increase in subsequent cohorts are 0.08, 0.16, and 0.32 mg/kg. Decision to proceed to the next higher dose cohort will be based upon a safety review of the included participants. Treatment will continue until intolerable toxicity or as per patient preference.

ELIGIBILITY:
Inclusion Criteria:

1. Huntington's Disease patients who Completed Study ER2001-001（NCT06024265）.
2. Patient has documented ability to understand the written study informed consent forms (ICFs) at the time of screening and has provided signed written informed consent prior to any study procedures.
3. HTT gene expansion testing with the presence of ≥40 CAG repeats.
4. Ability to undergo and tolerate MRI scans.
5. Ability to undergo and tolerate lumbar puncture.
6. All HD medications given for motor, behavioral, and cognitive symptoms have been stable for 3 months prior to Screening.
7. Other concomitant medications have been stable for 1 month prior to Screening.
8. organ function measured prior to administration of study treatment.
9. Postmenopausal or evidence of non-childbearing status for women of childbearing potential. Male patients must use a condom during treatment and for 6 months after the last dose of ER2001 when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception if they are of childbearing potential.

Exclusion Criteria:

1. History of attempted suicide or suicidal ideation with plan (i.e., active suicidal ideation) that required hospital visit and/or change in level of care within 12 months prior to screening.
2. Current active psychosis, confusional state, or violent behavior.
3. Bleeding tendency or history of coagulation disorder; As long as the investigator confirms that there is no evidence of bleeding tendency or coagulation dysfunction at present.
4. ECG with corrected QT interval (QTc) > 480 ms and/or indication of uncontrolled cardiac conditions, as judged by the investigator (e.g. unstable ischemia, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction,congestive heart failure, electrolyte disturbances, etc.)
5. Patients with HIV, Treponema pallidum, Hepatitis B, or Hepatitis C infection.
6. Need to take antiretroviral drugs, including antiretroviral drugs as preventive treatment.
7. Current or recurrent disease, infection, or other significant concurrent medical condition or medications that could confound clinical and laboratory evaluations or could affect a subject's safety or their ability to undergo the neurosurgical procedure or comply with the procedures and study visit schedule.
8. Clinical diagnosis of chronic migraines.
9. Presence of an implanted deep brain stimulation device, ventriculoperitoneal or other CSF shunt, or other implanted catheter.
10. Preexisting structural brain lesions (such as tumor, arteriovenous malformation) as assessed by a centrally read MRI scan during the screening period.
11. History of gene therapy, RNA or DNA investigational agents, such as antisense oligonucleotides (ASO), cell transplantation or any other experimental brain surgery.
12. Treatment with investigational therapy within 4 weeks prior to screening or 5 drug elimination half-lives of investigational therapy, whichever is longer.
13. Unable or unsafe to perform lumbar puncture on the patient.
14. In the Investigator's judgment, that Parkinson's disease, multiple system atrophy and other dystonia diseases may be combined.
15. Patients who are hypersensitive to any ingredients in the formulation of ER2001.
16. Malignancy within 5 years of screening, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated.
17. Concurrent or planned concurrent participation in any interventional clinical study, including explicit pharmacological and non- pharmacological interventions. Observational studies are acceptable.
18. Any serious medical condition or clinically significant laboratory, vital signs, or abnormalities at screening that, in the Investigator's judgment, precludes the patient's safe participation in and completion of the study.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of adverse events (AEs) and serious adverse events (SAEs) | Approximately 4.5 months
  To evaluate the safety and tolerability of ER2001 injection.

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | Approximately 4.5 months
  To assess the Pharmacokinetics (PK) of ER2001 injection.
Terminal half-life (t1/2) | Approximately 4.5 months
  To assess the Pharmacokinetics (PK) of ER2001 injection.
Area under the plasma concentration versus time curve from time 0 to the last quantifiable concentration (AUC0-t) | Approximately 4.5 months
  To assess the Pharmacokinetics (PK) of ER2001 injection.
Maximum concentration (Cmax) in cerebrospinal fluid (CSF) | Approximately 4.5 months
  To assess the Pharmacokinetics (PK) of ER2001 injection.

OTHER OUTCOMES:
Immunogenicity | Approximately 4.5 months
  To collect the incidence of Anti-Drug Antibodies (ADAs).
Change from baseline in the concentration of mutant huntingtin (mHTT) protein in cerebrospinal fluid (CSF) | Approximately 4.5 months
  To assess the dose-response relationship of ER2001 injection on mHTT protein change from baseline in cerebrospinal fluid (CSF).
Change from baseline in Unified Huntington's Disease Rating Scale (UHDRS) Total Functional Capacity (TFC) score | Approximately 4.5 months
  UHDRS is a research tool developed by Huntington Disease (HD) Study Group to provide a uniform assessment of the clinical features and course of HD. The UHDRS TFC comprises 5 functional domains associated with disability (occupation, finances, domestic chores, activities of daily living, and care level), with scores on each item ranging from 0 to either 2 or 3. The TFC total score is the sum of the 5 TFC items and can range from 0 to 13, with greater scores indicating higher functioning. Negative change from baseline indicates worsening.
Change from baseline in Unified Huntington's Disease Rating Scale (UHDRS) Total Motor Score (TMS) score. | Approximately 4.5 months
  UHDRS is a research tool developed by Huntington Disease (HD) Study Group to provide a uniform assessment of the clinical features and course of HD. The UHDRS TMS assesses all the motor features of HD and includes maximal chorea, maximal dystonia, ocular pursuit, saccade initiation and velocity, dysarthria, tongue protrusion, finger tapping, hand pronation and supination, luria, rigidity, bradykinesia, gait, tandem walking, and retropulsion pull test. Each of these was rated on a scale of 0 (normal motor function) to 4 (severely impaired motor function). TMS score is a sum of individual scores ranging from 0 (normal motor function) to 124 (severely impaired motor function). Lower TMS scores indicate better motor function.

CONTACTS AND LOCATIONS:
Overall Officials: pingyi xu, Ph.D, Principal Investigator — First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China